CLINICAL TRIAL: NCT03922841
Title: Pleural Disease: Phenotypes, Diagnostic Yield and Outcomes
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/2125
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Pleural Diseases
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with pleural disease: The subject must meet all of the following inclusion criteria to participate in this study.
  1. Evidence of pleural disease on chest radiograph or bedside ultrasound or Computed Tomography regardless of underlying aetiology
  2. No age or gender restrictions
  3. Ability to provide informed consent
  Interventions: Other: Pleural disease management

INTERVENTIONS:
Other: Pleural disease management — History, physical examination, pleural drainage, lab/radiographic investigations

SUMMARY:
Pleural disease i.e. with effusions or pneumothorax have a high disease burden to patients. This is because most patients require diagnostic and therapeutic interventions in the form of drainage and biopsies. With increasing age, the incidence of pleural disease is likely to rise with concomitant rise in pulmonary malignancy and infection.

The impact of pleural disease, especially ambulatory drainage depends not only on patient factors such as effusion size, cardiopulmonary co-morbidities and underlying aetiology. It also depends on socioeconomic factors such as ability to afford ambulatory equipment (which is not covered by Medisave), availability of care-givers and coping mechanisms.

To phenotype patients presenting to Singapore General Hospital with pleural disease and evaluate impact on outcomes of pleural interventions

This study will collect existing or prospective data that is part of standard clinical care

* Source of the data: electronic medical record of patients (ambulatory and inpatient)
* Data will be collected prospectively.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE

   Pleural disease i.e. with effusions or pneumothorax have a high disease burden to patients. This is because most patients require diagnostic and therapeutic interventions in the form of drainage and biopsies. With increasing age, the incidence of pleural disease is likely to rise with concomitant rise in pulmonary malignancy and infection.

   The impact of pleural disease, especially ambulatory drainage depends not only on patient factors such as effusion size, cardiopulmonary co-morbidities and underlying aetiology. It also depends on socioeconomic factors such as ability to afford ambulatory equipment (which is not covered by Medisave), availability of care-givers and coping mechanisms.

   Therefore, translating internationally accepted pleural interventions into an Asian context, moreover a Singaporean one, is challenging.
2. HYPOTHESIS AND OBJECTIVES

   Asian patients with pleural disease have unique phenotypes and outcomes from pleural interventions

   To phenotype patients presenting to Singapore General Hospital with pleural disease and evaluate impact on outcomes of pleural interventions
3. EXPECTED RISKS AND BENEFITS

   There are likely to be no benefits to subjects. They will not be subject to any novel therapy and their clinical data will only be collected.

   Risks are minimal because patients are subject to only standard therapy and existing clinical data collected. There will be no new additional interventions, consultations or hospital visits. They will be asked to complete validated quality of life surveys that will be included into the clinical record.
4. STUDY POPULATION

   4.1. List the number and nature of subjects to be enrolled.

   Patients will only be enrolled from those who present to Singapore General Hospital (either in an ambulatory or inpatient setting). There is no exclusion of women, children or minorities, although clinical catchment includes mostly adult patients.

   4.2. Criteria for Recruitment and Recruitment Process

   Subjects will be recruited if they already have radiographic evidence of pleural disease.

   4.3. Inclusion Criteria

   The subject must meet all of the following inclusion criteria to participate in this study.
   1. Evidence of pleural disease on chest radiograph or bedside ultrasound or Computed Tomography regardless of underlying aetiology
   2. No age or gender restrictions
   3. Ability to provide informed consent

   4.4. Exclusion Criteria Subjects who no radiographic evidence of pleural disease or who are unwilling/unable to provide informed consent
5. STUDY DESIGN AND PROCEDURES/METHODOLOGY

   This study will collect existing or prospective data that is part of standard clinical care
   * Source of the data: electronic medical record of patients (ambulatory and inpatient)
   * Data will be collected prospectively.
   * Time period: March 2018-2023
   * When subject collection is complete, the data will be de-identified and kept in an electronic database
   * Only principal investigator and co-investigators will have access to collected information.
   * Data be kept for 5 years after completion of study for data analysis and manuscript preparation
   * All electronic copies of data will be destroyed at the end of the study. All manual records if any will be shredded.

   Data that will be collected
   * Demographic data such as age, gender, ethnicity
   * Clinical data such as co-morbidities, medication history, American Society of Anaesthesiologists (ASA) status, smoking history, functional status (eg, ECOG)
   * Radiographic data including effusion size, septations, nodularity, underlying emphysema/fibrosis/consolidation/malignancy
   * Laboratory data: Serum and pleural LDH, glucose, albumin, total protein; Full blood counts, Renal panel, Liver Panel, Coagulation studies
   * Histopathology and microbiology results
   * Procedure (Pleural tap/catheter insertion/biopsy) details: designation of operator, procedure duration, anaesthesia used, complications, volume of effusion drained, number of biopsies taken, location of procedure, anti-microbials, pleurodesis.
   * Outcome measures such as radiographic improvement, duration of pleural catheter, quality of life using standardized measures (eg. St George's Respiratory Questionnaire), survival, hospital re-admission, further procedures needed (eg interventional radiology or thoracic surgery)

   Subjects may withdraw voluntarily from participation in the study at any time. They will have standard care as indicated by the managing physician
6. SAFETY MEASUREMENTS 6.1. Definitions

   An adverse event (AE) is any untoward medical occurrence that occurs as a result of the study. This will reported to CRIB.

   6.2. Collecting, Recording and Reporting of Adverse Events and Serious Adverse Events to CIRB

   PI will be responsible for submitting to the approving CIRB the completed serious AE Reporting Form within 7 calendar days after the investigator is aware of the event, followed by a complete report within 8 additional calendar days. AE that are related events should be reported at least annually (together with Study Status Report for annual review).

   6.3. Safety Monitoring Plan

   Not applicable. Current standard investigations and treatment to be provided to all subjects.

   6.4. Complaint Handling

   Complaints about the study will be escalated to the clinical Head of Department and included in reports to the CIRB.
7. DATA ANALYSIS

   7.1. Data Quality Assurance

   Data collection will be done by the investigators through the clinical team managing the patient to ensure completion and accuracy.

   7.2. Data Entry and Storage
   * Data will be entered and stored in a secure web application (REDCap)/password controlled hospital computer. When subject data collection is complete, the data will be de-identified and kept in an electronic database (password secured) for analysis. Only investigators will have access to the data.
   * There are no plans to keep any documentation of patients beyond the informed consent forms. These will be stored in the locked department office of the investigators.
8. SAMPLE SIZE AND STATISTICAL METHODS

   8.1. Determination of Sample Size

   The sample size is determined by the number of patients accrued into the database during the study period. As this is a non-comparative study, study size calculation not applicable.

   8.2. Statistical and Analytical Plans
   * Continuous safety analyses tracking for AE
   * Interim Analyses of data on an annual basis
9. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

   The CRIB will be permitted to audit the database as needed. Source documents are from electronic medical records.
10. QUALITY CONTROL AND QUALITY ASSURANCE

    Data collection will be done by the investigators through the clinical team managing the patient to ensure completion and accuracy.
11. ETHICAL CONSIDERATIONS

11.1. Informed Consent

Informed consent will be sought from the patient or legal guardian (in the case of minors) by the study investigators before any data collection is done.

11.2. Confidentiality of Data and Patient Records

* Data will be entered and stored in a secure web application (REDCap)/password controlled hospital computer. When subject data collection is complete, the data will be de-identified and kept in an electronic database (password secured) for analysis. Only investigators will have access to the data.
* There are no plans to keep any documentation of patients beyond the informed consent forms. These will be stored in the locked department office of the investigators.

ELIGIBILITY:
Inclusion Criteria:

* The subject must meet all of the following inclusion criteria to participate in this study.

  1. Evidence of pleural disease on chest radiograph or bedside ultrasound or Computed Tomography regardless of underlying aetiology
  2. No age or gender restrictions
  3. Ability to provide informed consent

Exclusion Criteria:

* Subjects who no radiographic evidence of pleural disease or who are unwilling/unable to provide informed consent

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited if they already have radiographic evidence of pleural disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Resolution of pleural disease | 30 days
  As above

CONTACTS AND LOCATIONS:
Overall Officials: Devanand Anantham, MRCP, Study Chair — Singhealth Foundation
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No data sharing involved